CLINICAL TRIAL: NCT00993525
Title: INTRAVITREAL RANIBIZUMAB FOR PERSISTENT NEW VESSELS IN DIABETIC RETINOPATHY (INIPE STUDY)
Brief Title: Intravitreal Ranibizumab For Persistent New Vessels In Diabetic Retinopathy(Inipe Study)
Acronym: INIPE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Apoio ao Ensino Pesquisa e Assitência do HCFMRPUSP (FAEPA) (Unknown); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Rodrigo Sanches Oliveira, Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3003/2009
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: diabetic retinopathy; ranibizumab; new vessels; intravitreal injection; Persistent retina new vessels
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravitreal anti-VEGF (Experimental): Intravitreal injection of 0.5 mg of ranibizumab
  Interventions: Drug: Intravitreal injection of ranibizumab

INTERVENTIONS:
Drug: Intravitreal injection of ranibizumab — 0.5 mg at week 0 0.5mg at weeks 12,24,36,48 if fluorescein leakage from active vessels on angiography
  Other Names: Lucentis

SUMMARY:
To evaluate the fluorescein angiographic and visual acuity effects of a single intravitreal injection of ranibizumab for the management of persistent new vessels associated with diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* persistent new vessels,defined as fine retinal vessels with dilated buds or tips covered with hemorrhage or associated with recurrent vitreous hemorrhage or paucity of accompanying fibrous tissue and/or increased in extent compared to previous visit,unresponsive to complete panretinal laser photocoagulation performed at least 4 months prior;
* logarithm of minimum angle of resolution (logMAR) best-corrected visual acuity of 0.17 (Snellen equivalent, 20/30) or worse.

Exclusion Criteria:

* history of vitrectomy in the study eye;
* history of thromboembolic event (including myocardial infarction or cerebral vascular accident);
* major surgery within the prior 6 months or planned within the next 28 days;
* uncontrolled hypertension;
* known coagulation abnormalities or current use of anticoagulative medication other than aspirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
total area of fluorescein leakage from active new vessels | baseline, weeks 1,6,12,24,36,48
Best corrected Visual Acuity (BCVA) | Baseline, weeks 1,6,12,24,36,48
central macular thickness | baseline, weeks 1,6,12,24,36,48

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Jorge, MD, Study Chair — University of Sao Paulo

REFERENCES:
- [Derived] Messias A, Ramos Filho JA, Messias K, Almeida FP, Costa RA, Scott IU, Gekeler F, Jorge R. Electroretinographic findings associated with panretinal photocoagulation (PRP) versus PRP plus intravitreal ranibizumab treatment for high-risk proliferative diabetic retinopathy. Doc Ophthalmol. 2012 Jun;124(3):225-36. doi: 10.1007/s10633-012-9322-5. Epub 2012 Mar 29. PMID 22457045